CLINICAL TRIAL: NCT00631670
Title: Stereotactic Body Radiation Therapy for Tumors Near the Spinal Cord
Brief Title: Stereotactic Body Radiation Therapy (SBRT) for Tumors Near the Spinal Cord
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 404-2005
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Results first posted 2012-01-25 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2010-06

CONDITIONS: Spinal Tumors
MeSH Terms: conditions — Spinal Cord Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Treatment Group (Experimental): 15 Gy dose in one stereotactic body radiation treatment
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- 25 Treatments Group (Experimental): 25 treatments, given once a day, Monday through Friday for about five weeks; Dose: 70 Gy at 2.8 Gy/treatment
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — 15 Gy in one treatment
  Arms: Single Treatment Group
Radiation: Stereotactic Body Radiation Therapy — Dose: 70 Gy at 2.8 Gy/treatment
  Arms: 25 Treatments Group

SUMMARY:
The purpose of this research study is to determine if Stereotactic Body Radiation Therapy (SBRT) is a good way to treat tumors near the spinal cord. Patients will either receive a single treatment or 25 days of treatment given once-a-day, Monday through Friday for about 5 continuous weeks. Our protocol uses life expectancy, patient preference, and tumor size to determine whether SBRT is delivered with 1 or 25 treatments. The single treatment dose is 15 Gy. The 25 treatment group is 70 Gy at 2.8 Gy/treatment.

DETAILED DESCRIPTION:
This protocol is a study of the use of Stereotactic Body Radiation Therapy (SBRT) for all types of primary or metastatic tumors near the spinal cord. The major goal of this study is to evaluate the efficacy and toxicity of a specific SBRT program in a prospective manner. The main outcome variables in this study are pain and neurologic function.

A major issue in delivering SBRT is the number of treatment sessions. There are advantages and disadvantages to both single and multi treatment programs. In this protocol, patients are offered SBRT with either a single treatment or 25 treatment days. This study is not designed to compare different SBRT schedules. A single treatment program is more convenient and likely to relieve symptoms sooner than a multi-session program. A program with 25 treatments may produce better long-term results. Our protocol uses life expectancy, patient preference, and tumor size to determine whether SBRT is delivered with 1 or 25 treatments.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in this protocol
* Patient of all ages are eligible
* All tumor types are eligible
* Patients with prior spine radiotherapy and/or surgery to the involved area are eligible
* The tumor target must be visible on MRI or CT scan
* Stereotactic Body Radiation Therapy (SBRT) on this protocol may produce a better outcome than conventional radiotherapy

Exclusion Criteria:

* Patients who are likely to have a satisfactory outcome with surgical resection, embolization, or radiofrequency ablation without the addition of radiotherapy
* Tumor size, shape, or location is such that it is not reasonable to think the patient may benefit from SBRT as given in this protocol
* The full extent of the tumor cannot be visualized on MRI or CT scan
* Delaying radiotherapy for the time that it takes to start SBRT may compromise outcome compared to starting conventional radiotherapy immediately
* The patient cannot be positioned reproducibly due to pain or other factors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-10; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amdur, MD, Principal Investigator — University of Florida- Radiation Oncology
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Treatment Group: 15 Gy dose of radiation in one treatment. Patients were offered the option of which arm they wished to participate in.
- 25 Treatments Group: 25 treatments, given once a day, Monday through Friday for about five weeks; Dose: 70 Gy at 2.8 Gy/treatment. Patients were offered the option to participate in which arm they preferred.
Period: Overall Study
Arm/Group | Single Treatment Group | 25 Treatments Group
Started | 21 | 0
Completed | 21 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Treatment Group | 25 Treatments Group | Total
Number analyzed (Participants) | 21 | 0 | 21
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 13 |  | 13
  >=65 years | 8 |  | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 58.5 (15.9) |  | 58.5 (15.9)
Gender [Number; unit: participants]
  Female | 9 |  | 9
  Male | 12 |  | 12
Region of Enrollment [Number; unit: participants]
  United States | 21 |  | 21

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Toxicities were graded using the RTOG-EORTC (Radiation Therapy Oncology Group-European Organization for Research and Treatment of Cancer) system and a descriptive system with which we coded any complication as mild, moderate, or severe based on our informal assessment of the complication's effect on overall quality of life. We assessed toxicity as "acute" meaning during treatment and "late" meaning several months after treatment ended.
Time Frame: 2 yrs
Measure: Number; unit: participants
Groups:
- Single Treatment Group: 15 Gy dose in one radiation treatment
Arm/Group | Single Treatment Group | 25 Treatments Group
Number analyzed (Participants) | 21 | 0
participants
  mild acute toxicity | 14 |
  moderate acute toxicity | 0 |
  severe acute toxicity | 0 |
  Late toxicity | 0 |

2. Secondary Outcome: Local Control
Description: Number of tumor sites with no evidence of progression of tumor at the site of radiosurgery
Time Frame: 1 year
Measure: Number; unit: tumors
Units Other Than Participants: tumors
Groups:
- Single Treatment Group: 15 Gy dose in one treatment
- 25 Treatments Grouop: 25 treatments, given once a day, Monday through Friday for about five weeks; Dose: 70 Gy at 2.8 Gy/treatment
Arm/Group | Single Treatment Group | 25 Treatments Grouop
Number analyzed (Participants) | 21 | 0
Number analyzed (tumors) | 25 | 0
tumors | 24 |

3. Secondary Outcome: Neurologic Function
Description: Number of patients with a change in neurological function of those who presented with a neurologic deficit from tumor compression. The McCormack score was noted for each patient and the interval change was determined informally as no neurological deficit, better, worse, or unchanged as noted below.
Time Frame: 2 years
Population: 6 patients presented with tumor-related deficits before treatment.
Measure: Number; unit: participants
Arm/Group | Single Treatment Group | 25 Treatments Group
Number analyzed (Participants) | 6 | 0
participants
  improved neurologic function | 0 |
  unchanged neurologic function | 6 |
  worse neurologic function | 0 |

4. Secondary Outcome: Pain Relief
Description: Number of patients who reported pain at baseline and reported experienced relief after treatment. Pain was defined on a 10 point scale with 0 being no pain and 10 being worst pain imaginable. Pain relief is defined as reporting a lower level of pain than that reported at baseline.
Time Frame: 12 weeks
Population: Patients who reported pain at baseline
Measure: Number; unit: participants
Arm/Group | Single Treatment Group | 25 Treatments Group
Number analyzed (Participants) | 14 | 0
participants | 6 |

5. Secondary Outcome: Overall One Year Survival
Description: Number of patients alive at one year after treatment
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Single Treatment Group | 25 Treatments Group
Number analyzed (Participants) | 21 | 0
participants | 5 |

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Single Treatment Group | 25 Treatments Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/0
Other Adverse Events (participants affected / at risk) | 14/21 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Treatment Group (N=21) | 25 Treatments Group (N=0)
Grade 1 Nausea (Gastrointestinal disorders) | 9 (9) | 0
Grade 2 Pharyngitis (Gastrointestinal disorders) | 5 (5) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes